CLINICAL TRIAL: NCT04028128
Title: Effects of Chronic Intake of High in Flavonols Cocoa on Body Composition, Adipokines and Exercise Performance
Brief Title: High Flavonols Cocoa Intake for the Improvement of Body Fat Composition in Athletes
Acronym: COCOFAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Mar Larrosa, Tenure Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AGL2016-77288-R-2
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Healthy Subjects
Keywords: Nutritional Supplement; High in flavanoids cocoa; Body Fat composition; Physical Exercise performance

STUDY DESIGN:
Intervention Model Description: Placebo controlled study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Cocoa and maltodextrin (placebo) are provided in identical sachets which are identified with the letters A and B respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocoa group (Experimental): The cocoa was provided in 5 g sachets. The intervention last 10 weeks. Cocoa was provided in a single daily dose of 5 g, which provided 425 mg of flavonoids
  Interventions: Dietary Supplement: Cocoa group
- Placebo group (Placebo Comparator): Maltodextrin (5 g) was supplied as placebo in sachets identical to those provided for cocoa.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Cocoa group — Athletes performed a training program and consumed 5 g of cocoa (425 mg of flavonoids) mixed with semi-skimmed fat milk, daily for 10 weeks.
  Arms: Cocoa group
Dietary Supplement: Placebo group — The athletes performed the same training program of the cocoa group and they took for 10 weeks 5 g of maltodextrin mixed with semi-skimmed fat milk.
  Arms: Placebo group

SUMMARY:
The decrease in body fat percentage improves exercise performance, reducing race time. The intake of cocoa improves the body fat composition in obese and diabetic people by improving their cardiovascular disease risk factors. Although epidemiological studies indicate that healthy subjects who consume cocoa have lower body fat composition, there is no study indicating whether cocoa improves fat composition in athletes. The aim of the study was to determine if the intake of cocoa rich in flavonoids improves the fat composition of athletes, modifying the systemic levels of adipokines (folistatin, myostatin and leptin), resulting in an improvement of physical performance.

DETAILED DESCRIPTION:
The objective of this project was to investigate the effects of chronic daily consumption of high in flavanols cocoa in body composition and performance of endurance athletes:

A randomized, blinded, parallel placebo controlled intervention study was carried out in endurance athletes . The number of male athletes enrolled in the study was 40, with ages between 18 and 50 years and an aerobic power consumption of oxygen greater than or equal to 55 mL / kg / min). The intervention was carried out for 10 weeks. Cocoa or placebo (maltodextrin) were supplied in sachets of a single daily dose. Cocoa provided 425 mg of flavanols/ day.

Athlete's body composition was evaluated by dual-energy X-ray absorptiometry (DEXA). Exercise performance was evaluated with a treadmill test protocol determining the maximum aerobic capacity and also by determining the time necessary to run a kilometer at maximum speed.

Adipokines (follistatin, myostatin and leptin) in plasma and serum samples were determined by ELISA.

Diet was determined by three 24h-recall questionnaries and a Food Frecuency questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Men.
* Age between 18 and 50 years
* Aerobic power of oxygen consumption greater than or equal to 55 mL / kg / min

Exclusion Criteria:

* Intake of chronical medication.
* Intake any type of nutritional or ergogenic supplements.
* Vegetarian or vegan diet
* Smoke.
* Any diagnosed disease at the time of inclusion or during the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — High performance sportsmen
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change of body fat mass at 10 weeks | Fat mass was analyzed at the beginning (baseline time = 0) and after 10 weeks of intervention
  Energy X-ray absorptiometry (DEXA).

SECONDARY OUTCOMES:
Change of lean mass at 10 weeks | Lean mass was analyzed at the beginning (baseline time) and after 10 weeks of intervention
  Energy X-ray absorptiometry (DEXA).
Change in Sport performance test at 10 weeks | Sport performance was analyzed at the beginning (baseline time) and after 10 weeks of intervention
  Assessment of maximal aerobic capacity by treadmill test
Change in Sport performance test 2 at 10 weeks | Sport performance was analyzed at the beginning (baseline time and after 10 weeks of intervention
  Measurement of the time that the sportsmen spend running one kilometer at the maximum speed.
Change from baseline of adipokines at 10 weeks | Myostatin and Follistatin were analyzed at the beginning and at the end of the 10-week intervention.
  Myostatin and Follistatin levels were measured in plasma
Change from baseline of leptin | Leptin was analyzed at the beginning and at the end of the 10-week intervention.
  leptin levels were measured in plasma by ELISA
Change in Dietary habits at 10 weeks | Diet was analyzed at the beginning (baseline dose) and after 10 weeks of intervention.
  Food Frequency Questionnaire. Consumption data were obtained for 93 foods. These data were entered into the DietSource software 3.0 (Novartis, Barcelona, Spain) to transform food data into percentage of carbohydrates, percentage of proteins and percentage of fat in the diet.
Change in Dietary habits 2 at 10 weeks | Diet was analyzed at the beginning (baseline dose) and after 10 weeks of intervention.
  24h recall questionnaire. This questionnaire was carried out 3 times on different days (2 weekdays and one weekend day) at the beginning (baseline) and after 10 weeks of intervention.These data were entered into the DietSource software 3.0 (Novartis, Barcelona, Spain) to transform food data into percentage of carbohydrates, percentage of proteins and percentage of fat in the diet.

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Larrosa Pérez, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Jose Ángel García Merino, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No